CLINICAL TRIAL: NCT07238582
Title: Effectiveness of an Innovative Chest Stabilizer in the Treatment of Rib Fractures: Impact on Respiratory Function, Complications, and Clinical Outcomes
Brief Title: Effectiveness of an Innovative Chest Stabilizer in Rib Fracture Treatment: Impact on Respiratory Function, Complications, and Clinical Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caner İşevi, MD (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Sponsor-Investigator, Caner İşevi, MD, Principal Investigator, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.ODM.0.20.08/ 715-779
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Rib Fractures; Blunt Chest Trauma; Thoracic Injuries; Pulmonary Complications
MeSH Terms: conditions — Rib Fractures; Thoracic Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: standard analgesic treatment or innovative chest stabilizer application.
Who Masked: Participant
Masking Description: Participants will not be informed about whether they receive standard treatment alone or the innovative chest stabilizer in addition to standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Analgesic Treatment (Active Comparator): Participants in this arm will receive standard pain management for rib fractures according to institutional clinical protocols. Treatment may include non-opioid or opioid analgesics, muscle relaxants, and supportive respiratory measures as clinically indicated. No chest stabilizer device will be applied.
  Interventions: Other: Standard Analgesic Therapy
- Innovative Chest Stabilizer (Experimental): Participants in this arm will receive standard analgesic treatment plus an innovative, non-invasive chest stabilizer. The stabilizer will be applied on the day of admission and used continuously for 10 days. Standard care includes routine analgesic medications administered according to institutional protocols. The chest stabilizer is designed to reduce pain, improve chest wall support, enhance respiratory mechanics, and potentially decrease pulmonary complications such as pneumonia or atelectasis.
  Interventions: Other: Standard Analgesic Therapy; Device: Innovative Chest Stabilizer

INTERVENTIONS:
Other: Standard Analgesic Therapy — Standard analgesic therapy provided according to institutional protocols for the management of rib fracture-related pain. Treatment may include routinely administered non-opioid or opioid analgesics and supportive respiratory care as clinically indicated. No chest stabilizer device is used in this intervention. This represents the standard of care and serves as the comparator for the study.
Device: Innovative Chest Stabilizer — A non-invasive chest wall stabilizing device applied on the day of hospital admission and used continuously for 10 days. The device is designed to reduce pain, improve chest wall support, enhance respiratory mechanics, and help prevent pulmonary complications such as pneumonia or atelectasis in patients with multiple rib fractures. The device is applied externally and does not require surgical intervention.
  Other Names: Non-Invasive Chest Wall Stabilizer
  Arms: Innovative Chest Stabilizer

SUMMARY:
This study aims to evaluate the effectiveness of an innovative, non-invasive chest stabilizer in patients with multiple rib fractures caused by blunt chest trauma. Rib fractures often lead to severe pain, breathing difficulties, and complications such as pneumonia or atelectasis. Participants will be randomly assigned to one of two groups: standard pain management or the new chest stabilizer, which will be used for 10 days.

The study will assess improvements in pain levels, breathing function (including FVC, FEV1, and PEF), and the occurrence of lung-related complications. Additional outcomes such as hospital stay, patient comfort, and skin reactions related to the device will also be evaluated. The goal of this research is to determine whether the innovative stabilizer can provide safer, more comfortable, and more effective treatment compared with current standard care for rib fracture patients.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 80 years. Blunt chest trauma with at least three rib fractures confirmed by imaging. Numeric Rating Scale (NRS) pain score ≥ 5 at rest, during deep inspiration, or with movement.

Able to perform spirometry reliably (FVC, FEV1, PEF). Hemodynamically stable and medically suitable for participation. Able and willing to provide informed consent.

Exclusion Criteria:

Age younger than 18 or older than 80 years. Penetrating chest trauma. Patients who have undergone surgical rib fixation. Active pneumonia, clinically significant atelectasis, or severe pulmonary infection at admission.

Uncontrolled cardiovascular, renal, or hepatic disease. Severe cognitive impairment, psychiatric disorders, or inability to comply with study procedures.

Severe respiratory failure requiring invasive mechanical ventilation. Skin infection, open wounds, or dermatologic conditions preventing stabilizer application.

Coagulopathy or contraindications to external chest compression. Pregnancy. Refusal or inability to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale (NRS) Pain Score From Baseline to Day 10 | Baseline and Day 10
  Pain intensity will be assessed using the 0-10 Numeric Rating Scale (NRS). Participants will report their pain score at rest and during deep inspiration on the day of admission (baseline) and again on Day 10. The outcome is the change in NRS score from baseline to Day 10. A greater reduction in NRS score indicates improved pain control. This outcome evaluates the primary clinical effect of the innovative chest stabilizer compared with standard analgesic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Medical Faculty, Department of Thoracic Surgery, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data because the study data will be used only for the primary analysis within the research team. De-identified datasets may be shared in the future upon reasonable request and after appropriate ethics review.